CLINICAL TRIAL: NCT03572101
Title: Living With Colorectal Cancer: Patient and Caregiver Experience
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); Alberta Health services (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Partnership Against Cancer (Unknown); Alberta Cancer Foundation (Other); Cancer Care Ontario (Other); Action Dignity (Other); Government of Alberta (Other Government)
Responsible Party: Principal Investigator, Aynharan Sinnarajah, Assistant Professor, Division of Palliative Medicine, Department of Oncology, University of Calgary
Other Study IDs: 201706HRC-387297
Record Dates: First submitted 2018-05-11; First posted 2018-06-28 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; palliative care; patients; caregivers; quality of life
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Calgary Patient Cohort: Patients with advanced colorectal cancer who are recruited from Calgary, Canada before, during, and after an early palliative care pathway becomes the new standard of care in Calgary.
- Calgary Caregiver Cohort: Caregivers of patients with advanced colorectal cancer who are recruited from Calgary, Canada before, during, and after an early palliative care pathway becomes the new standard of care in Calgary.
- Edmonton Patient Cohort: Patients with advanced colorectal cancer who are recruited from Edmonton, Canada during the same time period (no palliative care pathway introduced).
- Edmonton Caregiver Cohort: Caregivers of patients with advanced colorectal cancer who are recruited from Edmonton, Canada during the same time period (no palliative care pathway introduced).

SUMMARY:
This observational study will gather outcome and experience data of patients living with advanced colorectal cancer and their caregivers. The primary objective is to measure how quality of life in this population changes over time (before, during, and after a palliative pathway becomes the new standard of care in Calgary, Alberta, Canada).

DETAILED DESCRIPTION:
1. Background and Rationale: Using palliative care early, e.g. concurrent with disease-modifying therapies or from the time of diagnosis of advanced cancer, enhances quality of life for patients and their families and is associated with lower healthcare resource costs at end-of-life. Despite the evidence that early use of palliative care benefits patients and the healthcare system, most patients are referred late in their disease (e.g. <2 months from death). Our health services struggle to systematically provide early and integrated palliative care, to meet the needs of the cancer population. In Calgary, Alberta, typical of other Canadian centres, 60% of patients with metastatic gastrointestinal (GI) cancers have a late (< 3 months from end of life) or no palliative care referral (i.e. no contact with any palliative care service/provider). This lack of timely and early palliative care is associated with aggressive cancer care in 50% of patients, as compared to 25% in those who received earlier palliative care.

   A Knowledge to Action (KTA) initiative called Palliative Care Early and Systematic (PaCES) has identified gaps in providing early and systematic palliative care to advanced colorectal cancer (aCRC) patients. To address these gaps, a comprehensive care pathway delivering early, systematic palliative care to aCRC patients in Alberta, Canada will be developed as a new standard of care. The pathway will be implemented first in Calgary, Alberta, with Edmonton, Alberta as control site, to allow for testing and refinement before dissemination to Edmonton and across Alberta. As a result of the development of this new care pathway, over the next 3 years changes are anticipated in the delivery of care for aCRC patients.
2. Research question and objectives: This observational study will gather outcome and experience data of patients living with advanced colorectal cancer and their caregivers. The primary objective is to measure how quality of life in this population changes over time (before, during, and after a palliative pathway is introduced as the new standard of care in Calgary, Alberta).
3. Methods: An observational cohort study with interrupted time series (ITS) data collection will allow us to assess secular trends, determine if there is evidence of serial dependencies in the monthly measures, and to compare measures following system changes in Calgary while observing the same measures over the same time periods in Edmonton. The primary outcome will be how does EQ5D5L (a standardized instrument for use as a measure of health outcome) change over time for patients and caregivers. Questionnaires will be administered to patients monthly for 10 months then every 3 months until the end of the study or death. Questionnaires for the caregiver will be at enrollment, 1 month, then every 3 months until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* All advanced colorectal cancer patients > 18 years of age with one or more of the following:

  i) Failed first-line chemotherapy (disease progression on imaging); ii) Unable to receive first-line chemotherapy; iii) High symptom need (any score on the Edmonton Symptom Assessment System Revised (ESASr) ≥ 7); iv) Surprise question: In the opinion of a healthcare provider, would not be surprised if the patient died in the next 12 months.
* Caregivers of patients who meet inclusion/exclusion criteria.

Exclusion Criteria:

• A participant deemed inappropriate by clinic staff to be approached for an outcomes study for any reason (for example, in crisis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All advanced colorectal cancer patients at the Cross Cancer Institute (Edmonton, Canada), Tom Baker Cancer Centre (Calgary, Canada) and Holy Cross Centre (Calgary) will be screened and invited by their oncology healthcare providers to join the patient outcome and experience data collection. A caregiver, identified by each enrolled patient, may be invited to participate. For the purposes of this study, caregivers are defined as family or friends who provide unpaid assistance with tasks such as transportation and person care. Advanced Colorectal Cancer (aCRC) is defined as primary or metastatic cancer that is unlikely to be cured, controlled, or put into remission with treatment.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life (EQ-5D-5L scores) | Patients: at enrollment, then monthly for 10 months, then every 3 months. Caregivers: at enrollment, 1 month, then every 3 months. All until death or end of data collection (31 Dec 2020), whichever came first.
  The EQ-5D-5L tool will be used to characterize changes in patients' and caregivers' quality of life scores (index score and individual dimension scores) over time (i.e. as patients near end of life) and between cohorts (i.e. patients/caregivers in Calgary vs. patients/caregivers in Edmonton).

SECONDARY OUTCOMES:
Edmonton Symptom Assessment System-Revised (ESAS-r) symptoms (pain, tiredness, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath, and wellbeing) | Patients: at enrollment and then monthly for 10 months, then every 3 months thereafter until death or end of data collection (31Dec2020), whichever came first.
  The ESAS-r measures pain, tiredness, drowsiness, nausea, appetite, shortness of breath, depression, anxiety, and well-being, rated on a 0-10 scale of severity where 0 represents absence of the symptom and 10 represents the worst possible severity. The ESAS-r will be used to characterize the most common patient-reported symptoms, as well as changes in symptom scores (individual symptom scores as well as total score out of 90) over time (i.e. as patients near end of life), and between cohorts (i.e. patients in Calgary vs. patients in Edmonton).
Preparedness for caregiving | Caregivers: at enrollment, 1 month, then every 3 months until death of patient or end of data collection (31Dec2020), whichever came first.
  The Preparedness for Caregiving Scale is a tool that assesses caregiver readiness for providing care to another person, including preparedness for taking care of physical needs, emotional needs, accessing services, handling the stress of caregiving, making caregiving activities pleasant, handling emergencies, accessing health care system information, and overall preparedness. Items are rated on a 0-4 scale where 0 represents Not at all prepared and 4 represents Very well prepared. The Preparedness for Caregiving Scale will be used to characterize changes in caregivers' preparedness for caregiving (total score out of 32) over time (i.e. as patients near end of life) and between cohorts (i.e. caregivers in Calgary vs. caregivers in Edmonton).
Degree of engagement in advance care planning conversations | Patients: at enrollment and then monthly for 10 months, then annually until death or end of data collection (31Dec2020), whichever came first.
  The "My Conversations" tool is a questionnaire that assesses engagement in advance care planning conversations. The number of advance care planning conversation elements that a patient reports having discussed with a healthcare provider is scored on a 0-4 scale where 0 means no conversation elements and 4 means all conversation elements were discussed. The My Conversations tool will be used to characterize changes in the number of advance care planning conversation elements discussed over time (i.e. as patients near end of life), and between cohorts (i.e. patients in Calgary vs. patients in Edmonton).
Patient-reported concerns (emotional, social/family/spiritual, practical, physical, mobility, nutrition, informational, other) | Patients: at enrollment and then monthly for 10 months, then every 3 months thereafter until death or end of data collection (31Dec2020), whichever came first.
  The Canadian Problem Checklist is a checklist of emotional, social/family/spiritual, practical, physical, mobility, nutrition, and informational concerns. The Canadian Problem Checklist will be used to characterize patient concerns over time (i.e. as patients near end of life), and between cohorts (i.e. patients in Calgary vs. patients in Edmonton).

OTHER OUTCOMES:
Overall level of support received by patients/caregivers from homecare, cancer centre, long term care, hospital and hospice services at end of life | 8 weeks post death
  A post-bereavement survey (Caregiver Voice) will be used to characterize caregivers' experiences of patient's end of life care

CONTACTS AND LOCATIONS:
Overall Officials: Aynharan Sinnarajah, MD,MPH,CCFP, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Holy Cross Centre, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT03572101/Prot_SAP_000.pdf